CLINICAL TRIAL: NCT00770952
Title: Effects of Pioglitazone in Combination With Glimepiride in Comparison to Glimepiride Monotherapy on Metabolic Control in Patients With Type 2 Diabetes Mellitus
Brief Title: Efficacy of Pioglitazone and Glimepiride Combination Therapy in Treating Subjects With Type 2 Diabetes Mellitus.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Medical Director, Takeda Pharma GmbH, Aachen (Germany)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATS K020; 2006-002271-41 (EudraCT Number); D-PIO-112 (Other: Takeda ID); U1111-1114-3221 (Registry Identifier: WHO)
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2010-07

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus, Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus, Lipoatrophic; Dyslipidemias | interventions — Pioglitazone; glimepiride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone 30 mg to 45 mg QD + Glimepiride 2 mg to 4 mg QD (Experimental)
  Interventions: Drug: Pioglitazone and Glimepiride
- Glimepiride 4 mg to 6 mg QD (Active Comparator)
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: Pioglitazone and Glimepiride — Pioglitazone 30 mg, tablets, orally, once daily and Glimepiride 2 mg, tablets, orally once daily for two weeks; increased to:
  Pioglitazone 30 mg, tablets, orally, once daily and Glimepiride 4 mg, tablets, orally, once daily for two weeks; increased to:
  Pioglitazone 45 mg, tablets, orally, once daily and Glimepiride 4 mg, orally, once daily for up to 20 weeks.
  Other Names: ACTOS®
  Arms: Pioglitazone 30 mg to 45 mg QD + Glimepiride 2 mg to 4 mg QD
Drug: Glimepiride — Pioglitazone placebo-matching tablets, orally, once daily and Glimepiride 4 mg, tablets, orally once daily for two weeks; increased to:
  Pioglitazone placebo-matching tablets, orally, once daily and Glimepiride 5 mg, tablets, orally once daily for two weeks; increased to:
  Pioglitazone placebo-matching tablets, orally, once daily and Glimepiride 6 mg, tablets, orally once daily for up to 20 weeks.
  Arms: Glimepiride 4 mg to 6 mg QD

SUMMARY:
The purpose of this study is to determine the effect of pioglitazone, once daily (QD), and glimepiride combination therapy compared to glimepiride monotherapy in subjects with Type 2 Diabetes.

DETAILED DESCRIPTION:
Tight glycemic control is mandatory for the prevention and treatment of vascular complications in patients suffering from diabetes mellitus. After onset of Type 2 Diabetes, patients are usually treated with diet along with or without different combinations of oral drugs. One first-line drug class are sulfonylurea drugs that are preferably provided to patients who are not obese. The mode of action of sulfonylurea drugs is to increase beta-cell secretion, but it could be shown that they lead to deterioration of the beta-cell secretion product over time, resulting in increased proinsulin secretion. Since proinsulin is an independent cardiovascular risk factor, recent publications have demonstrated an increased risk for cardiovascular events in patients treated with sulfonylurea drugs as compared to other treatment methods.

Combination therapy of sulfonylurea drugs with glitazones has been shown to counterbalance the effect of deteriorated beta-cell secretion and to improve insulin sensitivity and the levels of proinsulin, C-peptide and other laboratory surrogate markers for cardiovascular risk. Proving that the treatment of diabetic patients with higher doses of beta cytotropic agents can be avoided and beta-cell function can be preserved by using pioglitazone in combination with low dose sulfonylurea drugs, it will be possible to optimize the treatment of patients with type 2 diabetes who are not controlled efficiently by sulfonylurea drugs monotherapy.

In this study patients will be enrolled who are inefficiently treated with a Glimepiride monotherapy. Patients will be either randomized to a combinational therapy of Pioglitazone and Glimepiride or Glimepiride monotherapy. If possible, study medication will be up-titrated to maximal dosage levels in both treatment arms to observe maximal and comparable treatment effects. Stable effects on beta-cell function will be observed after 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes according to the American Diabetes Association Criteria.
* Treatment with Glimepiride monotherapy (1-3 mg per day) 3 months before entering the study.
* Glycosylated hemoglobin greater than 6.5%, but less than 8.5% and/ or fasting plasma glucose greater than 7 mmol/l within the last 4 weeks.
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.

Exclusion Criteria:

* Type 1 Diabetes mellitus.
* History of hypersensitivity to the study drugs or to drugs with similar chemical structures.
* Progressive fatal disease.
* History of drug or alcohol abuse during the last 5 years.
* More than one unexplained episode of severe hypoglycemia within 6 months prior to entering the study.
* A history of significant cardiovascular (New York Heart Association stage I - IV), respiratory, gastrointestinal, hepatic (alanine aminotransferase greater than 2.5 times the upper limit of the normal reference range), renal (serum creatinine greater than 1.8 mg/dl; glomerular filtration rate less than 40 ml/min as estimated by the Cockroft-Gault formula), neurological, psychiatric and/or hematological disease, history of macular edema.
* Blood donation within the last 30 days.
* Is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * CYP2C9 inductors
  * CYP2C9 inhibitors
  * rifampicin
  * fluconazole
  * drugs used for treating type 2 diabetes (insulin, insulin analogous compounds and oral antidiabetic drugs)
* Pretreatment with thiazolidinediones within the last 12 months.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2006-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Homeostatic Model Assessment - Beta cell. | Week: 24 or Final Visit beyond week 12.

SECONDARY OUTCOMES:
Change from Baseline in Glycosylated Hemoglobin. | Week: 24 or Final Visit beyond week 12.
Change from Baseline in oral glucose tolerance testing. | Week: 24 or Final Visit beyond week 12.
Change from Baseline in Insulin. | Week: 24 or Final Visit beyond week 12.
Change from Baseline in Proinsulin. | Week: 24 or Final Visit beyond week 12.
Change from Baseline in C-peptide. | Week: 24 or Final Visit beyond week 12.
Change from Baseline in High sensitivity C-Reactive Protein. | Week: 24 or Final Visit beyond week 12.
Change from Baseline in Adiponectin. | Week: 24 or Final Visit beyond week 12.
Change from Baseline in Homeostatic Model Assessment - Sensitivity. | Week: 24 or Final Visit beyond week 12.
Change from Baseline in Triglycerides | Week: 24 or Final Visit beyond week 12.
Change from Baseline in Low Density Lipoprotein-Cholesterol | Week: 24 or Final Visit beyond week 12.
Change from Baseline in High Density Lipoprotein-Cholesterol | Week: 24 or Final Visit beyond week 12.
Change from Baseline in Total Cholesterol | Week: 24 or Final Visit beyond week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Adviser Clinical Research, Study Director — Takeda Pharma Gmbh, Aachen (Germany)
Locations (17):
- Germany (17):
  - Villingen-Schwenningen, Baden-Wurttemberg
  - Aschaffenburg, Bavaria
  - Ingolstadt, Bavaria
  - Frankfurt am Main, Hesse
  - Frielendorf, Hesse
  - Rotenburg an der Fulda, Hesse
  - Hanover, Lower Saxony
  - Dortmund, North Rhine-Westphalia
  - Siegen, North Rhine-Westphalia
  - Kallstadt, Rhineland-Palatinate
  - Mainz, Rhineland-Palatinate
  - Mayen, Rhineland-Palatinate
  - Neuwied, Rhineland-Palatinate
  - Rhaunen, Rhineland-Palatinate
  - Friedrichsthal, Saarland
  - Meissen, Saxony
  - Berlin, State of Berlin

REFERENCES:
- See also: ACTOS® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI